CLINICAL TRIAL: NCT07212972
Title: Mineral and Bone Disorder in Chronic Kidney Disease: A Comparative Analysis of Hemodialysis and Peritoneal Dialysis Modalities
Brief Title: Mineral Bone Disorder in Dialysis
Acronym: MBDialysis
Status: Completed | Type: Observational
Sponsor: Çanakkale Onsekiz Mart University (Other)
Responsible Party: Principal Investigator, Şeyma Eroğlu, Dr., Çanakkale Onsekiz Mart University
Other Study IDs: TZ-B
Record Dates: First submitted 2025-10-02; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2022-05

CONDITIONS: Chronic Kidney Failure; Chronic Kidney Disease-Mineral and Bone Disorder; Dialysis; Hemodialysis
MeSH Terms: conditions — Kidney Failure, Chronic; Chronic Kidney Disease-Mineral and Bone Disorder | interventions — Renal Dialysis; Peritoneal Dialysis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- dialysis: 167 patients diagnosed with CKD and undergoing HD or PD were included in the study
  Interventions: Other: Hemodialysis or peritoneal Dialysis

INTERVENTIONS:
Other: Hemodialysis or peritoneal Dialysis — Hemodialysis or peritoneal Dialysis

SUMMARY:
This study was conducted with 167 dialysis patients at Erciyes University Faculty of Medicine, Department of Internal Medicine, Department of Nephrology, and Dialysis Unit, with the approval of the Ethics Committee of Erciyes University Medical Faculty (date: 25.09.2019, no: 2019/673).

Patients aged ≥18 years, undergoing dialysis treatment, and having available data on serum calcium, phosphorus, parathormone, albumin, hemoglobin, blood urea nitrogen (BUN), creatinine, and dialysate calcium levels within the last six months were included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years,
* Diagnosed with chronic kidney disease (CKD) and undergoing dialysis treatment (hemodialysis or peritoneal dialysis)
* Availability of laboratory results within the last 6 months: serum calcium, phosphorus, parathormone, albumin, hemoglobin, blood urea nitrogen (BUN), creatinine, and dialysate calcium
* Patient consent to participate

Exclusion Criteria:

* Age < 18 years
* Patients not on dialysis treatment
* Missing or incomplete laboratory data
* History of malignancy, acute infection, or other systemic diseases interfering with mineral and bone metabolism
* Patients who did not provide consent or could not complete the questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study was performed with dialysis patients from Erciyes University Hospital, Faculty of Medicine, Department of Internal Medicine, and Department of Nephrology, and Dialysis Unit
Sampling Method: Probability Sample
Enrollment: 167 (Actual)
Dates: Start 2019-09-25 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2020-06-20 (Actual)

PRIMARY OUTCOMES:
Blood values | At the enrollment
  Serum levels of calcium, phosphorus, parathyroid hormone, albumin, hemoglobin, BUN, creatinine, and dialysate calcium

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes University Hospital, Faculty of Medicine, Department of Internal Medicine, and Department of Nephrology, and Dialysis Unit, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
They can be request.